CLINICAL TRIAL: NCT00125996
Title: A Randomised Controlled Study to Assess the Acute and Chronic Effects of Intravenous Iron Supplementation in Anaemic and Non-Anaemic Iron Deficient Patients With Chronic Heart Failure
Brief Title: Effect of Intravenous Ferrous Sucrose on Exercise Capacity in Chronic Heart Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Heart and Lung Institute (Other)
Collaborators: Wexham Park Hospital (Other); 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FERRIC-HF; FERRIC-Hef1; RD010; 131/03L
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 2005-01

CONDITIONS: Chronic Heart Failure; Heart Diseases; Anemia, Iron-Deficiency
Keywords: ANAEMIA; Iron Deficiency
MeSH Terms: conditions — Heart Diseases; Anemia, Iron-Deficiency; Anemia; Iron Deficiencies | interventions — Ferric Oxide, Saccharated

INTERVENTIONS:
Drug: Venofer (intravenous iron sucrose)

SUMMARY:
This is a two-center, randomised, single-blind (physician), prospective, controlled study to assess the acute (8 weeks) and chronic (16 weeks) effects of intravenous (IV) iron sucrose supplementation in anaemic and non-anaemic iron deficient patients with chronic heart failure (CHF).

The hypotheses are:

* Treatment of anaemic and non-anaemic iron-deficient CHF patients with IV iron sucrose improves exercise capacity as measured by peak VO2.
* IV iron sucrose is safe and well tolerated in subjects with moderate to severe CHF.

DETAILED DESCRIPTION:
Study Phase and Design:

Prospective two-centre, randomized, controlled, open-label, observer-blinded, parallel-group study

Primary Objective:

To evaluate the effect of intravenous (IV) iron supplementation on exercise tolerance, as determined by peak VO2.

Secondary Objectives:

* To evaluate the effects of IV iron supplementation on exercise duration, left ventricular (LV) structure and function, symptom status (NYHA class, Minnesota Living with Heart Failure Questionnaire [MLHFQ], and subjective fatigue score), and haematological and biochemical (haemoglobin [Hb], haematocrit [Hct], iron status, N-BNP, cytokines and oxidative stress) indices.
* To evaluate the safety profile of IV iron in subjects with moderate to severe CHF.

Sample Size:

42 subjects (28 IV iron, 14 placebo); 50% anaemic and 50% non-anaemic

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years of age and have signed written informed consent
* Stable symptomatic CHF; NYHA III/IV and left ventricular ejection fraction (LVEF) ≤40%, or if NYHA II then LVEF must be ≤35%, as assessed within last 6 months using echocardiographic or magnetic resonance imaging techniques.
* On optimal conventional therapy for at least 4 weeks prior to recruitment and without dose changes for at least 2 weeks.
* Peak VO2 ≤ 18 ml/kg/min on modified Naughton protocol cardiopulmonary exercise testing.
* Mean of the 2 screening Hb concentrations (week-2 and week-1) < 12.5 g/dl (anaemic group, 50% of study population) or 12.5-14.0 g/dl (non-anaemic group, 50% of study population).
* Ferritin <100 µg/l or 100-300 µg/l with TSAT <20%.
* Normal red cell folate and vitamin B12 status (according to local lab reference range).
* Resting blood pressure ≤160/100 mmHg.

Exclusion Criteria:

* History of acquired iron overload; known haemochromatosis or first relatives with haemochromatosis; and allergic disorders (asthma, eczema, and anaphylactic reactions).
* Known hypersensitivity to parental iron preparations.
* Known active infection, bleeding, malignancy and haemolytic anaemia.
* History of chronic liver disease and/or alanine transaminase (ALT) or aspartate transaminase (AST) >3 times the upper limit of the normal range; chronic lung disease; myelodysplastic disorder; and known HIV/AIDS disease.
* Recipient of immunosuppressive therapy or renal dialysis.
* History of erythropoietin, IV or oral iron therapy, and blood transfusion in previous 30 days.
* Unstable angina pectoris, as judged by the investigator; severe uncorrected valvular disease or left ventricular outflow obstruction; obstructive cardiomyopathy; uncontrolled fast atrial fibrillation or flutter (heart rate >110 beats per minute [bpm]); uncontrolled symptomatic brady- or tachyarrhythmias.
* Musculoskeletal limitation that, in the judgement of the investigator, would impair cardiopulmonary exercise testing.
* Pregnant or breast-feeding
* Inability to comprehend study protocol
* Parallel participation in another clinical trial

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-07; Study Completion 2006-02

PRIMARY OUTCOMES:
Change in peak VO2 from baseline to week 18

SECONDARY OUTCOMES:
Change in cardiopulmonary exercise duration from baseline to week 18
Change in distance walked during 6 minute walk test from baseline to end of repletion phase in treatment group or week 8 in control group, and week 18
Change in left ventricular (LV) systolic and diastolic dimensions, and function from baseline to week 18
Change in symptom status (New York Heart Association [NYHA] class, Minnesota Living with Heart Failure Questionnaire [MLHFQ], visual analogue fatigue scale) from baseline to week 1,week 8, and week 18
Change in haematological and biochemical indices (Hb, Hct, iron status, N-BNP, cytokines and oxidative stress) from baseline to week 18
Number and incidence of adverse events
Changes in liver function tests and renal function tests
Changes in vital parameters

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Poole-Wilson, MD,FRCP, Principal Investigator — NHLI, Imperial College School of Medicine
Locations (2):
- 4th Military Clinical Hospital, Weigla 5, Wroclaw, Poland
- Wexham Park Hospital, Wexham Park, Slough, Berkshire, United Kingdom

REFERENCES:
- [Derived] Okonko DO, Grzeslo A, Witkowski T, Mandal AK, Slater RM, Roughton M, Foldes G, Thum T, Majda J, Banasiak W, Missouris CG, Poole-Wilson PA, Anker SD, Ponikowski P. Effect of intravenous iron sucrose on exercise tolerance in anemic and nonanemic patients with symptomatic chronic heart failure and iron deficiency FERRIC-HF: a randomized, controlled, observer-blinded trial. J Am Coll Cardiol. 2008 Jan 15;51(2):103-12. doi: 10.1016/j.jacc.2007.09.036. PMID 18191732